CLINICAL TRIAL: NCT04002479
Title: A Feasibility and Safety Study of Intratumoral Diffusing Alpha Radiation Emitters on Advanced Pancreatic Cancer
Brief Title: Alpha Radiation Emitters Device for the Treatment of Advanced Pancreatic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-PANC-101
Record Dates: First submitted 2019-06-16; First posted 2019-06-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer; Unresectable Pancreatic Cancer; Metastatic Pancreatic Cancer; Pancreatic Adenocarcinoma
Keywords: pancreatic cancer; Unresectable Pancreatic Cancer; Metastatic Pancreatic Cancer; Pancreatic Adenocarcinoma; Pancreas Neoplasm; Alpha radiation; Pancreas Cancer; Pancreas Metastases
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of radioactive sources [Ra-224 containing stainless-steel 316LVM tubes- (Alpha DaRT seeds)]. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is a prospective, single-center, open label, single arm study. The study is designed to evaluate the feasibility, safety and preliminary efficacy of intratumoral alpha radiation mediated treatment with Alpha DaRT seeds for the treatment of advanced pancreatic cancer.

The study will be comprised of a screening period, DaRT insertion visit, acute follow-up phase of 4-6 weeks and a long-term follow up phase of 24 months. The total duration of the study will be 24 months from the DaRT insertion procedure.

30 patients with advanced pancreatic cancer will be recruited by the investigational site.

Eligible patients who meet inclusion/exclusion criteria (as assessed during the screening period) will be invited to the site for the procedure of DaRT seeds insertion. The patients will be monitored for a period of 24 months post insertion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically proven locally advanced (Stage II or III) or metastatic (Stage IV) pancreatic, adenocarcinoma
* Inoperable pancreatic cancer due to at least one of the following: a) unresectability, b) metastatic disease, c) medically unfit for surgery
* ECOG performance status ≤ 2
* Measurable lesion per RECIST (version 1.1) criteria
* Maximum lesion of 4cm in the longest diameter (including primary tumor and regional lymph nodes)
* ≥ 18 years of age
* Estimated life expectancy of at least 12 weeks
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test
* Subjects are willing to sign an informed consent

Exclusion Criteria:

* Prior chemotherapy does not exclude the patient
* Prior abdominal radiation therapy
* Concomitant chemotherapy or immunotherapy
* Borderline resectable pancreatic cancer and medically fit for surgery
* Connective tissue disease (scleroderma, lupus)
* Patients with significant comorbidities that the treating physician deems may conflict with the endpoints of the study (e.g., poorly controlled autoimmune diseases, vasculitis, etc.)
* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT
* High probability of protocol non-compliance (in opinion of investigator)
* Patients not willing to sign an informed consent form
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility - DaRT seed placement | Day 0 (Day of insertion)
  Assessment of the DaRT seed placement within the tumor or less than 5 mm from the tumor using CT imaging on the day of DaRT insertion.
Safety - Adverse events | 3 months
  Assessment of the frequency, severity and causality of acute AEs and SAEs related to DaRT seeds insertion. AEs and SAEs will be assessed and graded according to Common Terminology and Criteria for Adverse Events (CTCAE) version 5.0
Safety - Adverse events | 3 to 24 months
  Assessment of the frequency, severity and causality of Late AEs and SAEs related to DaRT seeds insertion. AEs and SAEs will be assessed and graded according to Common Terminology and Criteria for Adverse Events (CTCAE) version 5.0. The follow up will be carried out by phone calls every 2 months during the time between 3 to 24 months after DaRT seeds insertion

SECONDARY OUTCOMES:
Efficiency - Short-term effect | 4-6 weeks after DaRT seeds insertion
  Assessment of the objective response rate (ORR) following DaRT seeds insertion using CT scan
Tissue damage evaluation | Day -14 to 60 days after insertion
  Measuring CA19-9 as a marker to tissue damage. Elevation during treatment, and reduction as a result of tumor ablation. Serum levels of CA 19-9 can be measured using chemiluminescent assay on an Unicel DxI 800 analyzer (BeckmanCoulter, Brea, CA, USA).
Efficiency - Long-term effect | 2 years following DaRT seeds insertion
  Assessment of the overall survival (OS) following DaRT seeds insertion
Stent durability | Day of DaRT insertion up to 24 months.
  Stent durability will be assessed by the time elapsed from DaRT insertion to the need for follow-up referral for ERCP for stent change due to tumor ingrowth
Change in quality of life: EORTC-QLQ-C30 | Day -14 to 60 days after insertion
  Assessment of patient reported health-related Quality of Life (QoL) outcomes after DaRT treatment, using QoL questionnaires EORTC-QLQ-C30 (version 3.0). Scale range in score from 0 (best) to 100(worst).
Change in quality of life: QLQ-PAN26 | Day -14 to 60 days after insertion
  Assessment of patient reported health-related Quality of Life (QoL) outcomes after DaRT treatment, using QoL questionnaires QLQ-PAN26. The module comprises 26 questions assessing pain, dietary changes, jaundice, altered bowel habit, emotional problems related to pancreatic cancer, and other symptoms (cachexia, indigestion, flatulence, dry mouth, taste changes).

CONTACTS AND LOCATIONS:
Overall Officials: David Donath, MD, Principal Investigator — Brachytherapy Service Centre Hospitalier de l'Université de Montreal; Corey Miller, MD, Principal Investigator — Division of Gastroenterology, Jewish General Hospital
Locations (2):
- Canada (2):
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec